CLINICAL TRIAL: NCT02440061
Title: Ghrelin Effect on Beta Cell Function in Health and Disease #2
Brief Title: Ghrelin and Beta Cell Function in Diabetes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This protocol was replaced with a different one and therefore discontinued.
Sponsor: Jenny Tong, MD, MPH (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Jenny Tong, MD, MPH, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00060865; R01DK097550 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Ghrelin; age, BMI, and gender matched controls
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Arginine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Group: Type 2 Diabetes Mellitus (T2DM) (Active Comparator): Subjects with Type 2 Diabetes Mellitus (T2DM). Subjects will receive AG and saline infusions, but the order of which they receive will be random and they will not be told which one they are receiving on each given visit. Arginine will be used at both study visits.
  Interventions: Drug: Synthetic human AG; Drug: Arginine; Drug: 0.9% saline solution
- Control Group (Active Comparator): Control group of healthy subjects. Subjects will receive AG and saline, but the order of which they receive will be random and they will not be told which one they are receiving on each given visit. Arginine will be used at both study visits.
  Interventions: Drug: Synthetic human AG; Drug: Arginine; Drug: 0.9% saline solution

INTERVENTIONS:
Drug: Synthetic human AG — Synthetic human AG (0.28 μg/kg) bolus over 1 minute followed by 2 μg/kg/hr continuous infusion for 4.5 hours.
Drug: Arginine — Arginine hydrochloride (5 g) intravenously over 45 seconds.
Drug: 0.9% saline solution — A continuous infusion of 0.9% saline solution (control) for 4.5 hours.

SUMMARY:
Ghrelin is a hormone naturally produced in the stomach and the gut. The purpose of this research study is to determine the role of this gut hormone in the regulation of insulin secretion from the pancreas and glucose disposal after we eat. The investigators hypothesize that ghrelin has an effect on the pancreas and on how our body handles glucose after we eat. The investigators will compare insulin secretion and glucose changes during meal ingestion while either acyl ghrelin (AG) or saline (salt solution) is being infused through your vein on separate study days. AG is a form of the ghrelin hormone that has a small modification to it that allows it to bind to a specific receptor. The investigators hypothesize that AG has an effect on how the body handles glucose after a meal. AG has been approved by the U.S. Food and Drug Administration (FDA) for human research only. This study will also involve the use of a medicine called arginine, which is a naturally occurring product and found in many nutritional supplements. Its use in this study is investigational. The use of arginine helps maximize insulin release from the pancreas so the investigators can better examine whether AG affects insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

T2DM study subjects to be considered for the study must meet the following inclusion criteria:

1. Established T2DM with good to moderate glycemic control
2. HbA1c < 8.5%
3. Diabetes treatment with metformin, sulfonylurea, thiazolidinediones or combination of these medications; with no use of insulin during the study period
4. BMI ≤ 45.0 kg/m2

Control study subjects will be matched for age- (± 2 years), BMI (± 1.5 kg/m2) and gender and must meet the following inclusion criteria:

1. HbA1c ≤ 5.7%
2. Fasting plasma glucose ≤ 95 mg/dL
3. BMI ≤ 45.0 kg/m2

Exclusion Criteria:

All subjects will be excluded for the following reasons:

1. History of myocardial infarction or arrhythmia within the past year, abnormal electrocardiogram (ECG) with evidence of ischemia or arrhythmia, history or symptoms of congestive heart failure
2. Uncontrolled hypertension
3. History or active liver or renal disease (AST or ALT >2x upper limits of normal, calculated glomerular filtration rate [eGFR] <60 at screening)
4. History of pituitary or adrenal disorders or neuroendocrine tumor
5. Anemia defined as hematocrit <33% at screening
6. Active cancer diagnosis or currently undergoing cancer treatment
7. History of anorexia nervosa or previous gastrointestinal tract surgery
8. Pregnancy or lactation

Control subjects will be excluded for the following reasons:

1. History or clinical evidence of impaired fasting glucose or impaired glucose tolerance on a 75 g OGTT, established diabetes mellitus, or taking medications prescribed for diabetes
2. Use of medications that alter insulin sensitivity (i.e. niacin, glucocorticoids, metformin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Postprandial insulin secretion (ISR-meal) | approximately 8 weeks
  Postprandial insulin secretion (ISR-meal) will be derived from plasma C-peptide concentrations during MTT (0-240 min) using deconvolution with population estimates of C-peptide clearance.
Index of β-cell sensitivity to glucose | approximately 8 weeks
  Index of β-cell sensitivity to glucose will be calculated as incremental insulin/glucose (I/G) AUC (ΔAUCI/G).
Whole body insulin sensitivity using the Matsuda Index | approximately 8 weeks
  The Matsuda Index is a well-known index of insulin sensitivity derived from several glucose and insulin values obtained during a mixed meal
β-cell function (DI-meal) | approximately 8 weeks
  β-cell function (DI-meal) will be calculated as ΔAUCI/G x Matsuda Index

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tong, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center For Living, Durham, North Carolina, United States